CLINICAL TRIAL: NCT03493997
Title: An Investigative, Randomized, Open, Pilot Study to Assess the Tolerability, Safety and Efficacy of HAcid/CS Intravesical Instillations Plus an Oral Combination of Curcumin,Quercetin, HA and CS in Prevention of Radiation Induced Cystitis
Brief Title: Multicentre International STudy for the Prevention With Ialuril® of Radio-induced Cystitis (MISTIC)
Acronym: MISTIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Study Group for Urogenital Diseases, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MISTIC
Record Dates: First submitted 2018-01-25; First posted 2018-04-11 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy+Ialuril®+Ialuril Soft Gels® (Experimental): Radiotherapy+Ialuril®+Ialuril Soft Gels®
  Interventions: Combination Product: Radiotherapy+IAluril®+Ialuril Soft Gels®
- Radiotherapy only (Active Comparator): Radiotherapy only
  Interventions: Radiation: Radiotherapy only

INTERVENTIONS:
Combination Product: Radiotherapy+IAluril®+Ialuril Soft Gels® — Radiotherapy+IAluril®+Ialuril Soft Gels®
  Arms: Radiotherapy+Ialuril®+Ialuril Soft Gels®
Radiation: Radiotherapy only — Radiotherapy only
  Arms: Radiotherapy only

SUMMARY:
The study is randomized and it will be conducted in the field of routine clinical practice. A total of 100 consecutive patients planned to receive radiotherapy for prostate cancer will be enrolled.

The patients will enter the study as controls (50 patients that won't receive any experimental IMP) or as treated-group (50 patients that will be also treated with the experimental IMPs, Ialuril® and Ialuril® Soft Gels) according to a predefined, centre-specific randomization.

DETAILED DESCRIPTION:
Radiotherapy will last for 6 weeks. During planning of treatment, regimen and average dose to the whole bladder will be recorded to assess the impact of EBRT on urinary symptoms.

The treated-group will receive also intravesical Ialuril® weekly for 6 weeks (in the 24 hours before every radiation therapy weekly schedule), plus oral treatment with Ialuril® Soft Gels capsules (1 capsule twice a day after meals, at a distance of 12 hours, for 12 weeks).

The control-group will receive radiotherapy only for 6 weeks.

The Primary Objective is to assess the tolerability and safety of HA-CS intravesical instillations (Ialuril®) plus an oral combination of curcumin, quercetin, HA and CS (Ialuril® Soft Gels) in male patients undergoing radiotherapy for prostate cancer The efficacy of the treatment will be evaluated at the end of the study once received all the crfs.

ELIGIBILITY:
Inclusion Criteria:

* Male patients planned to receive primary radiotherapy for prostate cancer.

Exclusion Criteria:

* Female patients
* Patients with a life expectancy of less than 24 months
* with radiological confirmed metastasis
* with documented urethral strictures
* undergoing chemotherapy
* who received brachytherapy
* who received chemo-radiotherapy for prostate cancer in the past
* previously treated with Bacillus Calmette-Guerin (BCG)
* with post-void residual (PVR) > 200ml
* with clinical evidence of bladder calculi
* with neurogenic bladder or neurologic disease at risk for neurogenic bladder
* suffering from any lower urinary infections (UTIs, tuberculosis)
* with unstable cardiovascular disease
* with Congestive Heart Failure (CHF)
* with current nitrate use
* with current anticoagulants use (i.e. warfarin, heparin, etc.)
* with clinically significant hepatobiliary or renal disease
* with history of significant CNS injuries within 6 months
* with any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Rate of patients | 12 months
  The rate of patients who stopped treatment with intravesical or oral Ialuril due to intollerance or adverse events

SECONDARY OUTCOMES:
comparative analysis of score between the two groups through ICIQ | 12 months
  comparative analysis of score between the two groups (active arm vs. no drug arm)following questionnaires scores.
  Questionnaires:
  • ICIQ-Male Lower Urinary Tract Symptoms (ICIQ-MLUTS) questionnaire and bladder diary - Scale: Never - Occasionally
  * Sometimes - Most of the time - All of the time
comparative analysis of score between the two groups through EPIC | 12 months
  comparative analysis of score between the two groups (active arm vs. no drug arm)following questionnaires scores.
  Expanded Prostate Cancer Index Composite (EPIC) - Urinary Domain Scale :From 1 to 5 ( 1 smallest, 5 highest)
comparative analysis of score of QOL | 12 months
  comparative analysis of score between the two groups (active arm vs. no drug arm)following questionnaires scores.
  EQ-5D-5L (QoL) -
  Scale:
  I am not anxious or depressed I am slightly anxious or depressed I am moderately anxious or depressed I am severely anxious or depressed I am extremely anxious or depressed
comparative analysis of score between the two groups through IPSS | 12 months
  comparative analysis of score between the two groups (active arm vs. no drug arm)following questionnaires scores.
  IPSS Scale: 0 to 5 (0 worst - 5 best)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo LAzzeri, MD, Study Director — Gruppo di Studio per le Malattie Urogenitali
Locations (7):
- Italy (3):
  - Ospedali Careggi, Florence
  - Università "Vita-Salute" San Raffaele, Milan
  - University of Palermo, Italy, Palermo
- Slovakia (2):
  - St. Cyril and Method University Hospital, Bratislava
  - Fakultná nemocnica s poliklinikou, Prešov
- Universidad Autónoma de Barcelona, Barcelona, Spain
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lips IM, Dehnad H, van Gils CH, Boeken Kruger AE, van der Heide UA, van Vulpen M. High-dose intensity-modulated radiotherapy for prostate cancer using daily fiducial marker-based position verification: acute and late toxicity in 331 patients. Radiat Oncol. 2008 May 21;3:15. doi: 10.1186/1748-717X-3-15. PMID 18495016
- [Background] Pavlidakey PG, MacLennan GT. Radiation cystitis. J Urol. 2009 Sep;182(3):1172-3. doi: 10.1016/j.juro.2009.06.034. Epub 2009 Jul 22. No abstract available. PMID 19625037
- [Background] Smit SG, Heyns CF. Management of radiation cystitis. Nat Rev Urol. 2010 Apr;7(4):206-14. doi: 10.1038/nrurol.2010.23. Epub 2010 Mar 9. PMID 20212517
- [Background] Antonakopoulos GN, Hicks RM, Berry RJ. The subcellular basis of damage to the human urinary bladder induced by irradiation. J Pathol. 1984 Jun;143(2):103-16. doi: 10.1002/path.1711430205. PMID 6737117
- [Background] Denham JW, Hauer-Jensen M. The radiotherapeutic injury--a complex 'wound'. Radiother Oncol. 2002 May;63(2):129-45. doi: 10.1016/s0167-8140(02)00060-9. PMID 12063002
- [Background] Hurst RE. Structure, function, and pathology of proteoglycans and glycosaminoglycans in the urinary tract. World J Urol. 1994;12(1):3-10. doi: 10.1007/BF00182044. PMID 8012413
- [Background] Lazzeri M, Montorsi F. The therapeutic challenge of "chronic cystitis": search well, work together, and gain results. Eur Urol. 2011 Jul;60(1):78-80. doi: 10.1016/j.eururo.2011.03.039. Epub 2011 Apr 1. No abstract available. PMID 21474233
- [Background] Damiano R, Quarto G, Bava I, Ucciero G, De Domenico R, Palumbo MI, Autorino R. Prevention of recurrent urinary tract infections by intravesical administration of hyaluronic acid and chondroitin sulphate: a placebo-controlled randomised trial. Eur Urol. 2011 Apr;59(4):645-51. doi: 10.1016/j.eururo.2010.12.039. Epub 2011 Jan 18. PMID 21272992
- [Background] De Vita D, Giordano S. Effectiveness of intravesical hyaluronic acid/chondroitin sulfate in recurrent bacterial cystitis: a randomized study. Int Urogynecol J. 2012 Dec;23(12):1707-13. doi: 10.1007/s00192-012-1794-z. Epub 2012 May 22. PMID 22614285
- [Background] Cervigni M, Sommariva M, Porru D, Ostardo E, Tenaglia R, Giammò A, et al. A randomized, open-label, multicentre study of efficacy and safety of intravesical hyaluronic acid and chondroitin sulfate (HA 1.6% and CS 2%) vs dimethyl sulfoxide (DMSO 50%) in women with Bladder Pain Syndrome/Interstitial Cystitis (BPS/IC). Eur Urol Suppl 2014;13(1):e464.
- [Background] Cervigni M, Van Kerrebroeck PE, Dinis Oliveira P, Tarricone R, Guzman SA. Glycosaminoglycan-Replenishment Therapy: rationale for use and current evidence. EMJ Urol. 2014;1:41-47.
- [Background] Nordling J. Bladder Pain Syndrome/ Interstitial Cystitis. Update in Europe. International Journal of Urology 2014;21(Supplement S1):A1-A11.
- [Background] Crew JP, Jephcott CR, Reynard JM. Radiation-induced haemorrhagic cystitis. Eur Urol. 2001 Aug;40(2):111-23. doi: 10.1159/000049760. PMID 11528186
- [Background] Cox JD, Stetz J, Pajak TF. Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1341-6. doi: 10.1016/0360-3016(95)00060-C. No abstract available. PMID 7713792
- [Background] Charlson M, Szatrowski TP, Peterson J, Gold J. Validation of a combined comorbidity index. J Clin Epidemiol. 1994 Nov;47(11):1245-51. doi: 10.1016/0895-4356(94)90129-5. PMID 7722560
- [Background] Droller MJ, Saral R, Santos G. Prevention of cyclophosphamide-induced hemorrhagic cystitis. Urology. 1982 Sep;20(3):256-8. doi: 10.1016/0090-4295(82)90633-1. PMID 7123717
- [Background] Wei JT, Dunn RL, Litwin MS, Sandler HM, Sanda MG. Development and validation of the expanded prostate cancer index composite (EPIC) for comprehensive assessment of health-related quality of life in men with prostate cancer. Urology. 2000 Dec 20;56(6):899-905. doi: 10.1016/s0090-4295(00)00858-x. PMID 11113727
- [Background] Hamilton K, Bennett NC, Purdie G, Herst PM. Standardized cranberry capsules for radiation cystitis in prostate cancer patients in New Zealand: a randomized double blinded, placebo controlled pilot study. Support Care Cancer. 2015 Jan;23(1):95-102. doi: 10.1007/s00520-014-2335-8. Epub 2014 Jul 4. PMID 24993395
- [Background] Mottet N, Bastian PJ, Bellmunt J, van den Bergh RCN, Bolla M, van Casteren NJ, et al. Guidelines on Prostate Cancer. Uroweb 2014.